CLINICAL TRIAL: NCT05637749
Title: Mechanisms of Flow Regulation in a Novel Digital Serious Game for Rehearsing Complex Medical Subjects
Brief Title: Flow Regulation in Medical Serious Games
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Sreenivasulu Reddy Mogali, Assistant Professor, Head of Anatomy, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-2022-739
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Serious Games; Psychological Flow; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Serious game intervention to be played as is, without facilitation.
  Interventions: Other: Medical serious game intervention (educational)
- Intervention (Active Comparator): Serious game intervention to be played with facilitator present in game environment.
  Interventions: Other: Medical serious game intervention (educational)

INTERVENTIONS:
Other: Medical serious game intervention (educational) — Medical serious game designed to facilitate the rehearsal of diabetes management knowledge. Players are presented with a colony of individuals, all of whom have some form of diabetes, and are tasked to manage food, insulin, and medication intake throughout the day. The intervention may be played with a facilitator.
  Arms: Intervention
Other: Medical serious game intervention (educational) — Medical serious game designed to facilitate the rehearsal of diabetes management knowledge. Players are presented with a colony of individuals, all of whom have some form of diabetes, and are tasked to manage food, insulin, and medication intake throughout the day. The intervention may be played alone.
  Arms: Control

SUMMARY:
The goal of this study is to access the effect of facilitation on amount of psychological Flow generated in medical students playing a medical serious game. Students will be randomly assigned to play a serious game designed to revise diabetes management knowledge with and without a facilitator and the amount of Flow experienced compared. They will then be invited to partake in a focus group discussion to elicit insights into the mechanism of action governing facilitator-induced Flow

DETAILED DESCRIPTION:
The prevalence of diabetes and their complications is set to increase in line with Singapore's aging population, and the increasing complexities of medicine have left healthcare professionals beyond endocrinology reduced time or interest to seek out clinical sources of rehearsal. Despite having been taught diabetes management, knowledge not practiced fades over time, and delays or errors wrought by uncertainties may result in preventable loss of life or limb. Additionally, while many digital products exist to assist diabetes patients and caregivers, few cater to busy healthcare professionals and fewer account for differing levels of competency amongst them.

To address these needs, the study proposes the development and feasibility testing of a simulation-based diabetes management digital game incorporating a feature allowing for a human facilitator to moderate and personalise the rehearsal activity with consideration for a learner's strength and weaknesses.

The proposed mixed methods study thus presents the following aims:

Feasibility examination of the developed game intervention as an appropriate rehearsal tool for medical students

Comparing the degree of Flow (a state of total cognitive immersion in an activity) experienced by students who play the intervention with and without a facilitator

Generation of preliminary training data to guide either the development of more refined interventions wherein formal training data may be collected, or the direct training of a machine intelligence to assume the place of the human facilitator Map, where possible, the structure of the mechanism of action governing the interaction of facilitation and Flow in rehearsal-based digital serious games The study aims to accomplish these aims by first conducting a two-arm superiority randomised control trial (RCT) comparing the Flow Short Scale (7-point Likert scale survey measuring Flow) scores and in-game game analytics, such as number of correct decisions and reaction times, between students assigned to the facilitated and non-facilitated conditions.

Following this, students assigned to both conditions will be either be invited to partake in a focus group discussion, or given an open-ended questionnaire structured to solicit their attitudes, perceptions, and opinions of the game that may reveal insights into the mechanism of action governing facilitator-induced Flow.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in M1 through to M5 of the MBBS program under LKCMedicine.

Exclusion Criteria:

* Students who have previously partaken in play testing of the intervention
* Students not enrolled in the Bachelor of Medicine and Bachelor of Surgery (MBBS) program under LKCMedicine

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Flow Short Scale (FSS) scores | Immediately upon conclusion of the game activity
  The FSS comprises 13 items on a 7-point Likert scale ranging from 1 ("not at all) to 7 ("very much"). It demonstrates good construct validity, psychometric properties, and a stable three-factor structure comprising fluency of performance, absorption by activity, and perceived importance or outcome importance of said activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Lee Kong Chian School of Medicine, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan JW, Tan G, Lian X, Chong DKS, Rajalingam P, Dalan R, Mogali SR. Impact of Facilitation on Cognitive Flow in a Novel Diabetes Management Rehearsal Game for Health Professions Education: Mixed Methods, Open-Label, Superiority Randomized Controlled Trial. JMIR Serious Games. 2024 Jul 17;12:e54703. doi: 10.2196/54703. PMID 38900700